CLINICAL TRIAL: NCT02440464
Title: Multicenter Phase II, Double-blind Placebo Controlled Trial of Maintenance Ixazomib After Allogeneic Hematopoietic Stem Cell Transplantation for High Risk Multiple Myeloma (BMT CTN 1302)
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation With Ixazomib for High Risk Multiple Myeloma (BMT CTN 1302)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMT CTN 1302; U01HL069294-05 (NIH)
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Results first posted 2022-01-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Allogeneic Transplant; Maintenance Therapy; Anti-Myeloma Agents; Hematologic Disorders
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases | interventions — fludarabine; fludarabine phosphate; Melphalan; Bortezomib; ixazomib; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixazomib Maintenance (Experimental): Allogeneic HSCT and Fludarabine/Melphalan/Bortezomib conditioning followed by Ixazomib maintenance
  Interventions: Procedure: Allogeneic HSCT; Drug: Fludarabine; Drug: Melphalan; Drug: Bortezomib; Drug: Ixazomib
- Placebo (Placebo Comparator): Allogeneic HSCT and Fludarabine/Melphalan/Bortezomib conditioning followed by placebo maintenance.
  Interventions: Procedure: Allogeneic HSCT; Drug: Fludarabine; Drug: Melphalan; Drug: Bortezomib; Drug: Placebo

INTERVENTIONS:
Procedure: Allogeneic HSCT — Eligible patients with a Human Leukocyte Antigen (HLA)-matched related or unrelated donor will undergo allogeneic hematopoietic stem cell transplant at Day 0. For GVHD prophylaxis, patients will be given Tacrolimus from Day -3 until at least 6 months following initiation, at an intravenous daily dose of 0.015 mg/kg. This will be combined with an intravenous administration of Methotrexate at 5 mg/m2 on Days +1, +3, +6, and +11.
  Other Names: Allogeneic hematopoietic stem cell transplant
Drug: Fludarabine — Patients will receive conditioning treatment before and after HSCT. Fludarabine will be given at 30 mg/m2 intravenously on Day -6 through Day -3.
  Other Names: Fludara
Drug: Melphalan — Melphalan will be given at 70 mg/m2 intravenously on Days -4 and -3.
  Other Names: Alkeran
Drug: Bortezomib — Bortezomib will be administered at 1.3 mg/m2 intravenously on Day -3.
  Other Names: Velcade®
Drug: Ixazomib — Between 60 and 120 days following HSCT, patients randomized to the experimental arm will receive Ixazomib maintenance. Maintenance will begin at 3-mg oral doses on Days 1, 8, and 15 of a 28-day cycle. This will increase to 4-mg doses on the same cycle schedule, following successful completion of 3 cycles at the previous dosage, for a total of 12 cycles.
  Other Names: MLN9708; Ninlaro
  Arms: Ixazomib Maintenance
Drug: Placebo — Between 60 and 120 days following HSCT, patients randomized to the control group will be given 3 mg of placebo orally on Days 1, 8, and 15 of a 28-day cycle. This will increase to 4-mg doses on the same cycle schedule following successful completion of 3 cycles of placebo maintenance at the 3-mg dose. This will continue for a total of 12 cycles.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This study is designed to compare progression-free survival (PFS) from randomization among patients randomized on the BMT CTN 1302 protocol, "Multicenter Phase II, Double-blind Placebo Controlled Trial of Maintenance Ixazomib after Allogeneic Hematopoietic Stem Cell Transplantation for High Risk Multiple Myeloma". It is hypothesized that Ixazomib maintenance therapy will result in improved PFS in patients with high-risk multiple myeloma following Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) compared to placebo.

DETAILED DESCRIPTION:
The study is designed as a Phase II, multi-center double-blind trial that randomizes patients with high risk Multiple Myeloma to Ixazomib maintenance or placebo 60-120 days after allogeneic HSCT. The primary objective of this randomized trial is to compare progression free survival from randomization as a time to event endpoint between patients randomized to Ixazomib maintenance or placebo. Secondary objectives are to describe for each treatment arm: rates of grade II-IV and III-IV Graft-Versus-Host-Disease (GVHD), chronic GVHD, best disease response rates, disease progression, transplant related mortality, overall survival, rates of Grade ≥ 3 toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0, incidence of infections, and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet one of the following disease criteria:

   a. Patients with high risk multiple myeloma in partial response (PR) or better with no prior progression and are ≤ 24.0 months after autologous hematopoietic cell transplantation (HCT) (single or planned tandem), or are ≤ 24.0 months after initiation of systemic anti-myeloma therapy for patients without prior autologous HCT; or

   i. High risk is defined by the presence of any one of the following detected at any time prior to enrollment: deletion of chromosome 13 by conventional cytogenetics, hypodiploidy, abnormality in chromosome 1(1q amplification or 1p deletion), t(4;14), t(14;16), t(14;20) or deletion of 17p by fluorescence in situ hybridization (FISH) or conventional karyotyping; high risk criteria based on commercially available gene expression profiling (GEP)

   b. Patients with high risk multiple myeloma (see criterion 2.a.i. above) in very good partial response (VGPR) or better with 1 prior progression which occurred ≤ 24.0 months after autologous HCT (single or planned tandem), or ≤ 24.0 months after initiation of systemic anti-myeloma therapy for patients without prior autologous HCT; or

   i. Patients with one prior progression without measurable monoclonal paraprotein at the time of disease progression or relapse (< 1.0 g/dl in serum or < 200 mg/24hrs in urine) may be considered to have met VGPR criteria if < 5% plasma cells in bone marrow and ≥ 90% decrease in the difference between involved and uninvolved free light chain (FLC) levels from baseline (time of progression/relapse).

   ii. In patients with immunoglobulin G (IgG) kappa multiple myeloma (MM) receiving daratumumab: International Myeloma Working Group criteria for VGPR may not be achieved since daratumumab is known to increase the IgG kappa spike. In such cases the FLC and marrow may be used to establish VGPR, as above, with prior approval from the protocol co-chairs.

   c. Patients with standard risk multiple myeloma in VGPR or better (see criteria 2.b.i. and 2.b.ii. above) at the time of enrollment with 1 prior progression ≤ 24.0 months from single or planned tandem autologous HCT; or d. Patients with primary plasma cell leukemia in VGPR or better with no prior disease progression and are ≤ 18.0 months after autologous HCT, or are ≤ 18.0 months after initiation of anti-myeloma therapy without prior autologous HCT.
2. Patients must have a related or unrelated peripheral blood stem cell donor that meet one of the following criteria:

   1. A sibling donor who is a 6/6 match at HLA-A and -B (intermediate or higher resolution) and -DR Beta 1 (DRB1) (at high resolution using DNA-based typing) and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation OR
   2. A related donor (other than sibling) who is a 8/8 match for HLA-A, -B, -C (at intermediate or higher resolution) and -DRB1 (at high resolution using DNA-based typing) and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation OR
   3. An unrelated donor who is an 8/8 match at HLA-A, -B, -C, and -DRB1 (at high resolution using DNA-based typing) and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation.
3. Cardiac function: Ejection fraction > 40%
4. Estimated creatinine clearance greater than 40 mL/minute (using the Cockcroft-Gault formula and actual body weight)
5. Pulmonary function: Diffusing capacity of the lung for carbon monoxide (DLCO) ≥ 40% (adjusted for hemoglobin) and forced expiratory volume in one second (FEV1) ≥ 50%
6. Liver function: total bilirubin < 2x the upper limit of normal and alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 2.5x the upper normal limit (Patients with Gilbert's Disease are permitted to exceed the defined bilirubin value of 2x the upper limit of normal, however measurements of direct bilirubin should be done to confirm this diagnosis).
7. Female subjects (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two (2) effective methods of contraception at the same time, or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception) through 90 days after the last dose of maintenance therapy (see Section 2.6.2 for definition of postmenopausal).
8. Male subjects (even if surgically sterilized) must agree to one of the following: practice effective barrier contraception (see Section 2.6.4.1 for list of barrier methods), or practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of from the time of signing the informed consent through 90 days after last dose of maintenance therapy.
9. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
10. Able to comply with the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Karnofsky Performance Score < 70%
2. Prior allogeneic HCT
3. Patient with purely non-secretory multiple myeloma [absence of monoclonal protein (M protein) in serum as measured by electrophoresis and immunofixation and the absence of Bence Jones protein in the urine defined by the use of conventional electrophoresis and immunofixation techniques and the absence of involved serum free light chain > 100 mg/L].
4. Planned pre-emptive/prophylactic administration of donor lymphocytes (as per section 2.5.2)
5. Central Nervous System (CNS) involvement with multiple myeloma defined as cerebrospinal fluid (CSF) positivity for plasma cells or a parenchymal CNS plasmacytoma
6. Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
7. Presence of fluid collection (ascites, pleural, or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated.
8. Patients seropositive for the human immunodeficiency virus (HIV).
9. Patient with active Hepatitis B or C determined by serology and/or nucleic acid amplification test (NAAT).
10. Patients with hypersensitivity to bortezomib, boron or mannitol.
11. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 (ixazomib) including difficulty swallowing.
12. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
13. Patients with ≥ grade 2 sensory peripheral neuropathy.
14. Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure (see Appendix D), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
15. Female patients who are lactating or pregnant
16. Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years, which is in remission, will be reviewed on a case-by-case basis by the Protocol Officer or one of the Protocol Chairs.
17. Patients with multi-organ involvement by amyloidosis or evidence of amyloidosis related organ dysfunction.
18. Failure to have fully recovered (i.e., no toxicities > Grade 1 by CTCAE version 4.0) from the reversible effects of prior chemotherapy.
19. Patient with serious medical of psychiatric illness likely to interfere with participation on this clinical study
20. Participation in clinical trials with other investigational agents not included in this trial, ≤ 14.0 days of enrollment on this trial and throughout its duration.
21. Patients who have received radiation therapy within 3 weeks before transplant. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
22. Patients unable or unwilling to adhere to the study assessment schedule.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-08; Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - BMT Northside, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Texas /MD Anderson CRC, Houston, Texas
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to the NIH Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Bashir Q, Nishihori T, Pasquini MC, Martens MJ, Wu J, Alsina M, Anasetti C, Brunstein C, Dawson P, Efebera Y, Gasparetto C, Geller N, Giralt S, Hall AC, Koreth J, McCarthy P, Scott E, Stadtmauer EA, Vesole DH, Hari P. A Multicenter Phase II, Double-Blind, Placebo-Controlled Trial of Maintenance Ixazomib After Allogeneic Transplantation for High-Risk Multiple Myeloma: Results of the Blood and Marrow Transplant Clinical Trials Network 1302 Trial. Transplant Cell Ther. 2023 Jun;29(6):358.e1-358.e7. doi: 10.1016/j.jtct.2022.07.007. Epub 2022 Jul 12. PMID 35840087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on August 17, 2015 and closed to accrual on September 14, 2018 with 57 participants enrolled from 15 participating centers in the United States.
Pre-assignment Details: Five enrolled participants were not transplanted and an additional 9 participants dropped out of the study prior to randomization for a total of 43 participants who received a transplant and proceeded to randomization. The reasons for no transplant include progression (n=2), toxicity (n=2) and withdrew from study (n=1). The reasons for dropout prior to randomization include death (n=5), progression (n=1), neuropathy (n=1), severe infection (n=1) and withdrew from study (n=1).
Groups:
- Ixazomib Maintenance: Allogeneic hematopoietic stem cell transplantation (HSCT) and Fludarabine/Melphalan/Bortezomib conditioning followed by Ixazomib maintenance
  Allogeneic HSCT: Eligible patients with a Human Leukocyte Antigen (HLA)-matched related or unrelated donor will undergo allogeneic hematopoietic stem cell transplant at Day 0. For graft-versus-host disease (GVHD) prophylaxis, patients will be given Tacrolimus from Day -3 until at least 6 months following initiation, at an intravenous daily dose of 0.015 mg/kg. This will be combined with an intravenous administration of Methotrexate at 5 mg/m2 on Days +1, +3, +6, and +11.
  Fludarabine: Patients will receive conditioning treatment before and after HSCT. Fludarabine will be given at 30 mg/m2 intravenously on Day -6 through Day -3.
  Melphalan: Melphalan will be given at 70 mg/m2 intravenously on Days -4 and -3.
  Bortezomib: Bortezomib will be administered at 1.3 mg/m2 intravenously on Day -3.
  Ixazomib: Between 60 and 120 days following HSCT, patients randomized to the experimental arm will receive Ixazomib maintenance. Maintenance will begin at 3-mg oral doses on Days 1, 8, and 15 of a 28-day cycle. This will increase to 4-mg doses on the same cycle schedule, following successful completion of 3 cycles at the previous dosage, for a total of 12 cycles.
Period: Overall Study
Arm/Group | Ixazomib Maintenance | Placebo
Started | 21 | 22
Completed | 18 | 20
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Participants who were transplanted and randomized are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixazomib Maintenance | Placebo | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Median (Full Range); unit: years] | 52.6 [35.3 to 63.9] | 57.5 [44.9 to 64.7] | 55.9 [35.3 to 64.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Disease Classification [Count of Participants; unit: Participants] — High risk multiple myeloma (MM) is defined as participants with any of the following chromosomal changes detected by fluorescence in situ hybridization (FISH): t(4;14), t(14;16), del (17p), and abnormalities of chromosome 1 (1q21 amplifications; 1p deletion); deletion 13 or hypodiploidy by cytogenetics.
  Participants
    High Risk Multiple Myeloma | 12 | 12 | 24
    Standard Risk Multiple Myeloma | 6 | 6 | 12
    Primary Plasma Cell Leukemia | 3 | 4 | 7
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    100 | 2 | 5 | 7
    90 | 12 | 9 | 21
    80 | 5 | 5 | 10
    70 | 2 | 3 | 5
Disease Response [Count of Participants; unit: Participants] — Measure Description: Very Good Partial Response (VGPR): Partial Response (PR), paraprotein decrease or >= 90% serum paraprotein decrease, and a 90% involved light chain decrease. PR: >= 50% serum monoclonal paraprotein decrease and 24 hr urinary monoclonal decrease, or >= 50% involved and uninvolved free light chain (FLC) decrease or a 50% decrease in involved FLC w/ 50% ratio decrease, or >= 50% BM plasma cells decrease, or >= 50% soft tissue plasmacytomas decrease. Stable Disease: none of above and no progression.
  Participants
    Very Good Partial Response (VGPR) | 9 | 8 | 17
    Partial Response (PR) | 10 | 9 | 19
    Stable Disease or Progression | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival
Description: The primary endpoint compares progression-free survival as a time to event endpoint from randomization between patients randomized to ixazomib and placebo maintenance in high risk multiple myeloma. Participants are considered a failure of the primary endpoint if they die or suffer from disease progression or if they initiate non-protocol anti-myeloma therapy. Disease progression was evaluated using the International Uniform Response Criteria. Participants must meet one of the criteria for disease progression specified in the protocol. The time to this event is the time from randomization to progression, death, or initiation of non-protocol anti myeloma therapy whichever comes first. The Kaplan-Meier estimator was used to estimate progression-free survival during the 2 year post-transplant follow-up period. Participants who were event-free at two years post-transplant are censored at that time.
Time Frame: 12 months and 21 months post-randomization
Population: All randomized participants were included in the primary endpoint analysis.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants
  12 Months Post-randomization | 65.3 [50.0 to 77.0] | 72.7 [58.4 to 82.8]
  21 Months Post-randomization | 55.3 [40.0 to 68.1] | 59.1 [44.5 to 71.1]
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in progression-free survival time post-randomization among randomized subjects receiving Ixazomib vs Placebo maintenance therapy during the 21 month period post-randomization. This was compared between treatment arms using a log rank test; Test type: Superiority; p = 1.0, Log Rank — Statistical significance was determined using a pre-specified one-sided threshold of 0.10

2. Secondary Outcome: Percentage of Participants With Acute GVHD (Grades III-IV)
Description: Cumulative incidences of grade III-IV acute GVHD were determined using the Aalen-Johansen estimator. Death prior to acute GVHD is treated as the competing risk. Cumulative incidences are compared between treatment arms using Gray's test. Grading of acute GVHD was derived by consensus grading per BMT Clinical Trials Network (CTN) manual of procedures (MOP). The acute GVHD algorithm calculates the grade based on the organ (skin, GI and liver) stage and etiology/biopsy reported on the weekly GVHD form. Grade I aGVHD is defined as Skin stage of 1-2 and stage 0 for both GI and liver organs. Grade II aGVHD is stage 3 of skin, or stage 1 of GI, or stage 1 of liver. Grade III is stage 2-4 for GI, or stage 2-3 of liver. Grade IV is stage 4 of skin, or stage 4 of liver. Grade 4 is the worst outcome.
Time Frame: 100 days post-randomization
Population: All randomized subjects were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants | 9.5 [2.2 to 23.4] | 0.0 [0 to 0]
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with acute grade III-IV GVHD between the Ixazomib and Placebo arms during 100 days post-randomization, with death prior to acute GVHD treated as a competing risk. Cumulative incidences are compared between treatment arms using Gray's test; Test type: Superiority; p = 1.0, Gray's Test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05

3. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: Cumulative incidences of chronic GVHD were determined using the Aalen-Johansen estimator. Death prior to chronic GVHD is treated as the competing risk. Cumulative incidences are compared between treatment arms using Gray's test. Data of chronic GVHD were collected from providers and chart review according to the recommendations of the 2014 NIH Consensus Criteria. Eight organs are scored on a 0-3 scale to reflect degree of chronic GVHD involvement; 3 indicates the worst symptom. Liver and pulmonary function test results and use of systemic therapy for treatment of chronic GVHD are also recorded.
Time Frame: 12 months and 21 months post-randomization
Population: All randomized participants were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants
  12 Months Post-randomization | 68.6 [46.8 to 82.9] | 63.6 [43.3 to 78.3]
  21 Months Post-randomization | 68.6 [46.8 to 82.9] | 63.6 [43.3 to 78.3]
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with chronic GVHD between the Ixazomib and Placebo arms during 21 months post-randomization, with death prior to chronic GVHD treated as a competing risk. Cumulative incidences are compared between treatment arms using Gray's test; Test type: Superiority; p = 1.0, Gray's Test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05

4. Secondary Outcome: Percentage of Participants With Best Response to Treatment After Randomization
Description: Response was assessed using the International Uniform Response Criteria. Best response is the best of all the disease response status at each assessment time point after randomization. The order from best to worst is: Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD). All disease classifications are relative to the patient's disease status prior to allogeneic transplant (i.e. study entry). This outcome was compared between treatment groups using all response data up to 2 years post-transplant. These response data were summarized separately for patients in sCR/CR at the time of randomization vs. those who were not in sCR/CR at the time of randomization. Within each group (in sCR/CR vs not in sCR/CR at randomization), best response to treatment was compared between treatment groups using a Fisher's Exact test instead of a chi-square test because of the small sample size.
Time Frame: 2 years post-transplant
Population: All randomized participants were included in the analysis. Participants were divided into those in sCR/CR at the time of randomization vs. those who were not in sCR/CR at the time of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
Participants
  Participants in sCR/CR at Randomization: number analyzed (Participants) | 9 | 11
  Participants in sCR/CR at Randomization: Stringent Complete Response (sCR) | 6 | 5
  Participants in sCR/CR at Randomization: Complete Response (CR) | 2 | 4
  Participants in sCR/CR at Randomization: Very Good Partial Response (VGPR) | 0 | 1
  Participants in sCR/CR at Randomization: Partial Response (PR) | 0 | 0
  Participants in sCR/CR at Randomization: Stable Disease (SD) | 0 | 0
  Participants in sCR/CR at Randomization: Progressive Disease (PD) | 1 | 1
  Participants Not in sCR/CR at Randomization: number analyzed (Participants) | 12 | 11
  Participants Not in sCR/CR at Randomization: Stringent Complete Response (sCR) | 3 | 4
  Participants Not in sCR/CR at Randomization: Complete Response (CR) | 2 | 3
  Participants Not in sCR/CR at Randomization: Very Good Partial Response (VGPR) | 4 | 4
  Participants Not in sCR/CR at Randomization: Partial Response (PR) | 2 | 0
  Participants Not in sCR/CR at Randomization: Stable Disease (SD) | 0 | 0
  Participants Not in sCR/CR at Randomization: Progressive Disease (PD) | 1 | 0
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; Participants in sCR/CR at Randomization; Test type: Superiority — The null hypothesis is that there is no difference in the proportions of participants in the best response to treatment categories between the Ixazomib and Placebo arms during 2 years post-transplant among participants in sCR/CR at randomization. These proportions were compared using Fisher's Exact test; p = 0.890, Fisher Exact; Statistical significance was determined using a pre-specified one-sided threshold of 0.05
Statistical Analysis 2: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants in the best response to treatment categories between the Ixazomib and Placebo arms during 2 years post-transplant among participants not in sCR/CR at randomization. These proportions were compared using Fisher's Exact test; Test type: Superiority; p = 0.754, Fisher Exact — Statistical significance was determined using a pre-specified one-sided threshold of 0.05

5. Secondary Outcome: Percentage of Participants With Response to Treatment
Description: Response was assessed using the International Uniform Response Criteria. All disease classifications are relative to the patient's disease status prior to allogeneic transplant (i.e. study entry). Response to treatment after randomization (sCR, CR, VGPR, or PR) is summarized in each arm post-transplant at 18 months and 24 months post-transplant. These response data were summarized separately for patients in sCR/CR at the time of randomization vs. those who were not in sCR/CR at the time of randomization.
Time Frame: 18 months and 24 months post-transplant
Population: All randomized participants were included in the analysis. Participants were divided into those in sCR/CR at the time of randomization vs. those who were not in sCR/CR at the time of randomization. Reasons participants were not evaluable were either they withdrew from study or missed an assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
Participants
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: number analyzed (Participants) | 9 | 11
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: Stringent Complete Response (sCR) | 3 | 3
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: Complete Response (CR) | 2 | 3
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: Very Good Partial Response (VGPR) | 1 | 2
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: Partial Response (PR) | 0 | 0
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: Stable Disease (SD) | 0 | 0
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: Progressive Disease (PD) | 1 | 1
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: Died Before Evaluation | 1 | 2
  Response to Treatment at 18 Months Post-transplant for Participants in sCR/CR at Randomization: Not Evaluable | 1 | 0
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: number analyzed (Participants) | 12 | 11
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: Stringent Complete Response (sCR) | 2 | 3
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: Complete Response (CR) | 1 | 2
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: Very Good Partial Response (VGPR) | 3 | 4
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: Partial Response (PR) | 1 | 0
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: Stable Disease (SD) | 1 | 0
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: Progressive Disease (PD) | 0 | 0
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: Died Before Evaluation | 0 | 0
  Response to Treatment at 18 Months Post-transplant for Participants Not in sCR/CR at Randomization: Not Evaluable | 4 | 2
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: number analyzed (Participants) | 9 | 11
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: Stringent Complete Response (sCR) | 2 | 1
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: Complete Response (CR) | 3 | 6
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: Very Good Partial Response (VGPR) | 1 | 0
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: Partial Response (PR) | 0 | 0
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: Stable Disease (SD) | 0 | 0
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: Progressive Disease (PD) | 1 | 1
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: Died Before Evaluation | 1 | 2
  Response to Treatment at 24 Months Post-transplant for Participants in sCR/CR at Randomization: Not Evaluable | 1 | 1
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: number analyzed (Participants) | 12 | 11
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: Stringent Complete Response (sCR) | 2 | 2
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: Complete Response (CR) | 1 | 2
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: Very Good Partial Response (VGPR) | 3 | 4
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: Partial Response (PR) | 0 | 0
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: Stable Disease (SD) | 1 | 0
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: Progressive Disease (PD) | 0 | 0
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: Died Before Evaluation | 0 | 1
  Response to Treatment at 24 Months Post-transplant for Participants Not in sCR/CR at Randomization: Not Evaluable | 5 | 2

6. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Disease progression was evaluated using the International Uniform Response Criteria. Participants in sCR/CR must meet at least one of the criteria for disease progression specified in the protocol for sCR/CR participants; those not in sCR/CR must meet at least one of the disease progression criteria specified in the protocol for those not in sCR/CR. The cumulative incidence of progression from randomization will be estimated for each treatment arm using the Aalen-Johansen estimator, with death in remission treated as a competing risk. Initiation of anti-myeloma therapy will be considered evidence of progression. Participants who were event-free at two years post-transplant are censored at that time.
Time Frame: 12 months and 21 months post-randomization
Population: All randomized participants were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants
  12 Months Post-randomization | 34.7 [17.8 to 52.3] | 27.3 [13.0 to 43.8]
  21 Months Post-randomization | 44.7 [25.6 to 62.1] | 36.4 [19.8 to 53.3]
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with progression between the Ixazomib and Placebo arms during 21 months post-randomization, with death prior to progression treated as a competing risk. Cumulative incidences are compared between treatment arms using Gray's test; Test type: Superiority; p = 1.0, Gray's Test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05

7. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Overall survival (OS) is defined as freedom from death from any cause. OS post-randomization is estimated for each arm using the Kaplan-Meier estimator and compared between arms using the log rank test. Participants who are alive at two years post-transplant are censored at that time. Confidence intervals for values of 100% were not calculated and are shown as 100%.
Time Frame: 12 months and 21 months post-randomization
Population: All randomized participants are included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants
  12 Months Post-randomization | 100.0 [100.0 to 100.0] | 90.9 [73.7 to 97.1]
  21 Months Post-randomization | 94.7 [75.6 to 99.0] | 86.4 [68.4 to 94.5]
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in overall survival time post-randomization among randomized subjects receiving Ixazomib vs Placebo maintenance therapy during the 21 month period post-randomization. This was compared between treatment arms using a log rank test; Test type: Superiority; p = 0.174, Log Rank — Statistical significance was determined using a pre-specified one-sided threshold of 0.05

8. Secondary Outcome: Percentage of Participants With Treatment-Related Mortality (TRM)
Description: Treatment-related mortality is defined as death occurring in a patient from causes other than disease relapse or progression. The cumulative incidence of treatment-related mortality (TRM) post-randomization is estimated for each treatment arm using the Aalen-Johansen estimator, with progression treated as a competing risk. Participants who were event-free at two years post-transplant are censored at that time. Confidence intervals for values of 0% were not calculated.
Time Frame: 12 months and 21 months post-randomization
Population: All randomized participants were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants
  12 Months Post-randomization | 0 [NA to NA] — Because there were no events, the confidence interval was not calculated. | 0 [NA to NA] — Because there were no events, the confidence interval was not calculated.
  21 Months Post-randomization | 0 [NA to NA] — Because there were no events, the confidence interval was not calculated. | 4.5 [0.5 to 16.5]
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with treatment-related mortality between the Ixazomib and Placebo arms during 21 months post-randomization, with progression treated as a competing risk. Cumulative incidences are compared between treatment arms using Gray's test; Test type: Superiority; p = 0.173, Gray's Test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05

9. Secondary Outcome: Percentage of Participants With Toxicities Post-randomization by Toxicity Type
Description: Toxicities are graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. Higher grades correspond to worse symptoms with the minimum grade being a 0 and the maximum grade being a 5. Toxicities post-randomization are described for each treatment arm by the type of toxicity as well as peak overall grade.
Time Frame: 2 years post-randomization
Population: All randomized participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
Participants
  Maximum Toxicity Grade : 0 - 2 | 8 | 6
  Maximum Toxicity Grade : 3 | 13 | 14
  Maximum Toxicity Grade : 4 | 0 | 1
  Maximum Toxicity Grade : 5 | 0 | 1
  Abnormal Liver Symptoms | 3 | 2
  Dysgeusia | 1 | 2
  Encephalopathy | 0 | 0
  Grade 3-5 Allergic Reaction | 0 | 1
  Grade 3-5 Anaphylaxis | 0 | 0
  Grade 3-5 Blood/Lymphatic Toxicity | 5 | 8
  Grade 3-5 Cardiac Toxicity | 6 | 7
  Grade 3-5 Fatigue | 3 | 3
  Grade 3-5 Fever | 0 | 0
  Grade 3-5 GI Toxicity | 6 | 7
  Grade 3-5 Hearing Loss | 0 | 0
  Grade 3-5 Hemorrhage | 0 | 0
  Grade 3-5 Hepatobiliary/Pancreas | 1 | 7
  Grade 3-5 Hyperthyroidism | 0 | 0
  Grade 3-5 Hypothyroidism | 0 | 1
  Grade 3-5 Metabolic Toxicity | 4 | 6
  Grade 3-5 Musculoskeletal Toxicity | 1 | 3
  Grade 3-5 Nervous System Toxicity | 4 | 4
  Grade 3-5 Ocular Toxicity | 0 | 2
  Grade 3-5 Renal Toxicity | 0 | 5
  Grade 3-5 Respiratory Toxicity | 2 | 8
  Grade 3-5 Skin/Subcutaneous Tissue Toxicity | 1 | 5
  Grade 3-5 Vascular Toxicity | 2 | 3
  Hepatitis | 0 | 1
  Intestinal Obstruction | 1 | 0
  Liver Failure | 0 | 0
  Severe Muscle Weakness/Paralysis | 0 | 1
  Sudden Vision Loss | 0 | 0
  Tumor Lysis Syndrome | 1 | 0

10. Secondary Outcome: Percentage of Participants With Toxicities Post-randomization by Time Point
Description: Toxicities are graded using NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. Higher grades correspond to worse symptoms with the minimum grade being a 0 and the maximum grade being a 5. The cumulative incidence of Grade ≥ 3 toxicity was estimated at 6, 12 and 18 months post randomization using Aalen-Johansen estimators for each treatment group. Death from a cause other than toxicity was treated as a competing risk. Comparison of cumulative incidence between the two treatment arms was done using a Z test at fixed time points.
Time Frame: 6, 12 and 18 months post-randomization
Population: All randomized participants were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants
  6 Months Post-randomization | 57.1 [36.9 to 73.1] | 63.6 [43.4 to 78.3]
  12 Months Post-randomization | 61.9 [41.3 to 77.1] | 68.2 [47.7 to 82.0]
  18 Months Post-randomization | 61.9 [41.3 to 77.1] | 72.7 [52.1 to 85.6]
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with Grade 3-5 toxicities between the Ixazomib and Placebo arms during 6 months post-randomization, with death from a cause other than toxicity treated as a competing risk. Cumulative incidences are estimated at 6, 12 and 18 months post randomization using Aalen-Johansen estimators for each treatment group. Comparison of cumulative incidence between treatment arms was done using a Z test at fixed time points; Test type: Superiority; p = 0.258, Z test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05
Statistical Analysis 2: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with Grade 3-5 toxicities between the Ixazomib and Placebo arms during 12 months post-randomization, with death from a cause other than toxicity treated as a competing risk. Cumulative incidences are estimated at 6, 12 and 18 months post randomization using Aalen-Johansen estimators for each treatment group. Comparison of cumulative incidence between treatment arms was done using a Z test at fixed time points; Test type: Superiority; p = 0.252, Z test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05
Statistical Analysis 3: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with Grade 3-5 toxicities between the Ixazomib and Placebo arms during 18 months post-randomization, with death from a cause other than toxicity treated as a competing risk. Cumulative incidences are estimated at 6, 12 and 18 months post randomization using Aalen-Johansen estimators for each treatment group. Comparison of cumulative incidence between treatment arms was done using a Z test at fixed time points; Test type: Superiority; p = 0.258, Z test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05

11. Secondary Outcome: Percentage of Participants With Infections Post-randomization by Infection Type
Description: All Grade 2 and 3 infections are reported according to the BMT CTN MOP (Manual of Procedures) where a higher grade corresponds to more severe symptoms. The number of participants with post-randomization infections in each treatment arm is described by severity and type of infection.
Time Frame: 2 years post-randomization
Population: All randomized participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
Participants
  Participants with Infections | 8 | 11
  Maximum Severity: Grade 2 | 6 | 10
  Maximum Severity: Grade 3 | 2 | 1
  Participants with Bacterial Infection | 3 | 2
  Participants with Viral Infection | 6 | 11
  Participants with Fungal Infection | 0 | 1
  Participants with Other Infection | 1 | 0

12. Secondary Outcome: Percentage of Participants With Infections Post-randomization by Time Point
Description: All Grade 2 and 3 infections are reported according to the BMT CTN MOP (Manual of Procedures) where a higher grade corresponds to more severe symptoms. The cumulative incidence of severe, life-threatening, or fatal infections (Grade 3), treating death as a competing event, are estimated at 6, 12 and 18 months post randomization using Aalen-Johansen estimators for each treatment group. Comparison of cumulative incidence between the two treatment arms was done using a Z test at fixed time points.
Time Frame: 6, 12 and 18 months post-randomization
Population: All randomized participants were included in the analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
percentage of participants
  6 Months Post-randomization | 4.8 [0.6 to 17.0] | 0.0 [NA to NA] — Because there were no events, the confidence interval was not calculated.
  12 Months Post-randomization | 4.8 [0.6 to 17.0] | 0.0 [NA to NA] — Because there were no events, the confidence interval was not calculated.
  18 Months Post-randomization | 4.8 [0.6 to 17.0] | 0.2 [-10.6 to 11.1]
Statistical Analysis 1: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with Grade 3 infections between the Ixazomib and Placebo arms during 6 months post-randomization, with death from a cause other than infection treated as a competing risk. Cumulative incidences are estimated at 6, 12 and 18 months post randomization using Aalen-Johansen estimators for each treatment group. Comparison of cumulative incidence between treatment arms was done using a Z test at fixed time points; Test type: Superiority; p = 1.0, Z test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05
Statistical Analysis 2: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with Grade 3 infections between the Ixazomib and Placebo arms during 12 months post-randomization, with death from a cause other than infection treated as a competing risk. Cumulative incidences are estimated at 6, 12 and 18 months post randomization using Aalen-Johansen estimators for each treatment group. Comparison of cumulative incidence between treatment arms was done using a Z test at fixed time points; Test type: Superiority; p = 1.0, Z test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05
Statistical Analysis 3: Comparison: Ixazomib Maintenance vs Placebo; The null hypothesis is that there is no difference in the proportions of participants with Grade 3 infections between the Ixazomib and Placebo arms during 18 months post-randomization, with death from a cause other than infection treated as a competing risk. Cumulative incidences are estimated at 6, 12 and 18 months post randomization using Aalen-Johansen estimators for each treatment group. Comparison of cumulative incidence between treatment arms was done using a Z test at fixed time points; Test type: Superiority; p = 1.0, Z test — Statistical significance was determined using a pre-specified one-sided threshold of 0.05

13. Secondary Outcome: Functional Assessment of Cancer Therapy (FACT) - Bone Marrow Transplant (BMT) Total Score
Description: The FACT-BMT version 4.0 instrument is comprised of the Functional Assessment of Cancer Therapy - General (FACT-G), which evaluates the health-related quality of life (HQL) of patients receiving treatment for cancer, and the BMT Concerns module, that addresses disease and treatment-related questions specific to bone marrow transplant. This scale goes from 0 to 196 where higher scores indicate better functioning. The FACT-BMT Total, which has all items in the FACT-G and BMT modules, was used as the outcome measure. This self-reported questionnaire was completed at transplant, randomization, 6 months following the start of maintenance therapy (which corresponds to 6 months post-randomization), and 24 months post-transplant. Comparisons between treatment groups were performed prior to maintenance, 6 months post-randomization and at 24 months after transplant. Only English and Spanish speaking patients were eligible to participate in the quality of life component of this trial.
Time Frame: Randomization, 6-months post-randomization, 24 months post-transplant
Population: Randomized participants who completed the questionnaire are included.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale
  Randomization: number analyzed (Participants) | 19 | 21
  Randomization | 100.0 [61.2 to 148.0] | 110.0 [86.0 to 146.0]
  6 Months Post-randomization: number analyzed (Participants) | 16 | 11
  6 Months Post-randomization | 121.4 [58.5 to 148.0] | 114.0 [76.7 to 141.0]
  24 Months Post-transplant: number analyzed (Participants) | 12 | 9
  24 Months Post-transplant | 121.5 [72.5 to 147.0] | 109.0 [68.0 to 133.0]
  Change from Randomization to 6 Months Post-randomization: number analyzed (Participants) | 14 | 10
  Change from Randomization to 6 Months Post-randomization | 5.0 [-46.0 to 50.0] | 7.0 [-33.3 to 29.0]
  Change from Randomization to 24 Months Post-transplant: number analyzed (Participants) | 12 | 9
  Change from Randomization to 24 Months Post-transplant | 12.6 [-15.0 to 49.0] | 3.0 [-42.0 to 32.8]

14. Secondary Outcome: Medical Outcomes Study (MOS) - Short Form 36 (SF-36) Score
Description: The MOS SF-36 instrument is a general assessment of health quality of life with eight components: Physical Functioning, Role Physical, Pain Index, General Health Perceptions, Vitality, Social Functioning, Role Emotional, and Mental Health Index. The scale is 0 to 100 where 0 is maximum disability and 100 is no disability, so the higher the score the more positive the outcome. The Physical Component Summary (PCS) and Mental Component Summary (MCS) were used as the outcome measures in summarizing the SF-36 data for this study. This self-reported questionnaire was completed at transplant, randomization, 6 months following the start of maintenance therapy (which corresponds to 6 months post-randomization), and 24 months post-transplant. Comparisons between treatment groups were performed prior to maintenance, 6 months post-randomization and at 24 months after transplant. Only English and Spanish speaking patients were eligible to participate in the quality of life component of this trial.
Time Frame: Randomization, 6 months post-randomization, 24 months post-transplant
Population: Randomized participants who completed the questionnaire are included.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Ixazomib Maintenance | Placebo
Number analyzed (Participants) | 21 | 22
score on a scale
  PCS: Randomization: number analyzed (Participants) | 19 | 21
  PCS: Randomization | 38.7 [22.9 to 57.5] | 41.5 [22.8 to 55.0]
  PCS: 6 Months Post-randomization: number analyzed (Participants) | 17 | 12
  PCS: 6 Months Post-randomization | 47.9 [23.4 to 58.4] | 41.2 [23.3 to 58.6]
  PCS: 24 Months Post-transplant: number analyzed (Participants) | 12 | 9
  PCS: 24 Months Post-transplant | 45.1 [30.9 to 58.9] | 45.7 [36.6 to 58.5]
  PCS: Change from Randomization to 6 Months Post-randomization: number analyzed (Participants) | 15 | 11
  PCS: Change from Randomization to 6 Months Post-randomization | 3.3 [-3.7 to 22.4] | 1.0 [-15.7 to 12.1]
  PCS: Change from Randomization to 24 Months Post-transplant: number analyzed (Participants) | 12 | 9
  PCS: Change from Randomization to 24 Months Post-transplant | 4.7 [-19.8 to 29.4] | 7.8 [-10.4 to 19.4]
  MCS: Randomization: number analyzed (Participants) | 19 | 21
  MCS: Randomization | 51.5 [23.4 to 64.3] | 49.9 [37.7 to 63.3]
  MCS: 6 Months Post-randomization: number analyzed (Participants) | 17 | 12
  MCS: 6 Months Post-randomization | 54.8 [26.8 to 63.4] | 54.5 [43.2 to 60.8]
  MCS: 24 Months Post-transplant: number analyzed (Participants) | 12 | 9
  MCS: 24 Months Post-transplant | 56.1 [29.4 to 66.0] | 49.5 [22.8 to 58.5]
  MCS: Change from Randomization to 6 Months Post-randomization: number analyzed (Participants) | 15 | 11
  MCS: Change from Randomization to 6 Months Post-randomization | -0.6 [-18.1 to 16.7] | 5.3 [-10.6 to 8.2]
  MCS: Change from Randomization to 24 Months Post-transplant: number analyzed (Participants) | 12 | 9
  MCS: Change from Randomization to 24 Months Post-transplant | 4.9 [-7.5 to 16.6] | -2.5 [-32.0 to 11.0]

ADVERSE EVENTS:
Time Frame: 2 years post-randomization
Description: Adverse event (AE) reporting was done using the BMT CTN's Manual of Procedures (MOP). Unexpected, grade 3-5 AE were reported through an expedited AE reporting system. Expected AEs were reported using National Cancer Institute (NCI)'s Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 at regular intervals as defined on the Form Submission Schedule and reported in the secondary outcome "Toxicities". All fatal (Grade 5) expected adverse events were reported in an expedited manner.
Groups:
- Enrolled Not Randomized: Participants who enrolled in the study but were not randomized to treatment.
Arm/Group | Ixazomib Maintenance | Placebo | Enrolled Not Randomized
All-Cause Mortality (participants affected / at risk) | 1/21 | 3/22 | 5/14
Serious Adverse Events (participants affected / at risk) | 11/21 | 12/22 | 7/14
Other Adverse Events (participants affected / at risk) | 4/21 | 7/22 | 2/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib Maintenance (N=21) | Placebo (N=22) | Enrolled Not Randomized (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cryptitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Graft versus host disease (Immune system disorders) | 2 (2) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib Maintenance (N=21) | Placebo (N=22) | Enrolled Not Randomized (N=14)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02440464/Prot_SAP_ICF_000.pdf